CLINICAL TRIAL: NCT00177242
Title: Phase II Study of Gefitinib and Docetaxel as Salvage Therapy in Advanced Pancreatic Carcinoma
Brief Title: Study of Gefitinib and Docetaxel as Salvage Therapy in Advanced Pancreatic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Nathan Bahary, MD, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-027
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: pancreas; pancreatic
MeSH Terms: conditions — Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
This is a phase II, open-label trial of Gefitinib and docetaxel in patients having one prior regimen of chemotherapy for with metastatic pancreatic carcinoma.

DETAILED DESCRIPTION:
Initial therapy for metastatic pancreatic carcinoma is inadequate, and there is no effective second line therapy. Docetaxel has known single agent activity in pancreatic carcinoma, resulting in a median survival of 5.9 months, similar to gemcitabine, when assessed in Phase II studies (10) and pancreatic tumors are known to express EGFR. We propose that the combination of docetaxel with Gefitinib will have activity against pancreatic carcinoma, whether the regimen is administered as first or second-line therapy for metastatic disease. Given the toxicity profiles of both agents, we believe this will be a well-tolerated regimen. In fact, preliminary analysis of a phase II study of docetaxel and Gefitinib with an identical regimen in non-small cell lung cancer patients showed this regimen to be safe and active.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas that is surgically inoperable
* Must have had one prior chemotherapeutic regimen for advanced disease (Prior radiation with a radiation sensitizer for locally advanced disease or adjuvant therapy is not considered a prior regimen for purpose of this study)
* Disease must be measurable by RECIST criteria; measurable disease will be defined as at least one lesion that can be accurately measured in at least one dimension measuring at least 2 cm conventional CT or MRI or 1 cm with spiral CT scans (Appendix A)
* Aged 18 years or older
* ECOG performance status of 0 - 2 (see Appendix B)
* Able to take oral medications without difficulty
* Adequate bone marrow function as evidenced by an ANC > 1500/mL and platelet count > 100, 000/mL
* Adequate renal function as evidenced by serum creatinine within institutional limits or creatinine clearance > 60 ml/minute if above upper institutional limits (ULN)
* Adequate hepatic function as evidenced by ALT, AST, and total bilirubin within ULN. If hepatic metastases are present, ALT and AST may be up to 5 x ULN.
* Provision of written informed consent
* Men and women of childbearing potential must be willing to practice acceptable methods of birth control to prevent pregnancy. This is a precautionary measure for use of Gefitinib and docetaxel.

Exclusion Criteria:

* Known severe hypersensitivity to Gefitinib or docetaxel or any of the excipients of these products (i.e. polysorbate 80)
* Previous treatment with Gefitinib or docetaxel.
* Other coexisting malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma or squamous cell carcinoma of the skin or cervical cancer in situ.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's Wort
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment.
* Treatment with radiation therapy or chemotherapy within 28 days before Day 1 of trial treatment
* Any unresolved chronic toxicity greater then CTC grade 2 from previous anticancer therapy (except alopecia)
* Incomplete healing from previous oncologic or other major surgery.
* Pregnancy or breast feeding (women of childbearing potential).
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Ascertain the median survival of advanced pancreatic cancer patients treated with Gefitinib and docetaxel.

SECONDARY OUTCOMES:
Determine the response rate, time to disease progression, survival rate at 6- month intervals after treatment start, and safety profile of Gefitinib and docetaxel as treatment for advanced pancreatic cancer
Determine the time course of serial CA19-9 measurements during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Foon, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Ramanathan RK, Abbruzzese J, Dragovich T, Kirkpatrick L, Guillen JM, Baker AF, Pestano LA, Green S, Von Hoff DD. A randomized phase II study of PX-12, an inhibitor of thioredoxin in patients with advanced cancer of the pancreas following progression after a gemcitabine-containing combination. Cancer Chemother Pharmacol. 2011 Mar;67(3):503-9. doi: 10.1007/s00280-010-1343-8. Epub 2010 May 12. PMID 20461382